CLINICAL TRIAL: NCT01010828
Title: Efficacy and Safety of Vanguard PS Knee Joint System Using MIS Technique
Brief Title: Review on Minimally Invasive Skin Incision in Vanguard PS Artificial Knee Joint System
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Zimmer Biomet (Industry)
Collaborators: Biomet Japan, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: JP12
Record Dates: First submitted 2009-11-09; First posted 2009-11-10 (Estimated); Last update posted 2019-03-27 (Actual); Status verified 2019-03

CONDITIONS: Gonarthrosis Patients Who Need Artificial Knee Joint Total Replacement

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Tri-Vector Approach (Active Comparator)
  Interventions: Procedure: Incision technique
- Mini Mid-Vastus Approach (Experimental)
  Interventions: Procedure: Incision technique

INTERVENTIONS:
Procedure: Incision technique — Tri-Vector Approach retains the majority of 3 vectors of quadriceps.
  Arms: Tri-Vector Approach
Procedure: Incision technique — Mini Mid-Vastus Approach
  Arms: Mini Mid-Vastus Approach

SUMMARY:
This study will show whether Tri-Vector method can ensure more extensive visual field and conduct the precise surgery when compared with Mini Mid-Vastus method by conducting 2 types of skin incision approach, Tri-Vector for 36 patients or Mini-Mid Vastus for 36 patients in Vanguard PS artificial knee joint total replacement observational period before and during surgery.

ELIGIBILITY:
Inclusion Criteria:

* The patients who need artificial knee joint replacement in ordinary medical consultation are selected as the subjects.

Exclusion Criteria:

* Patients with infections such as osteomyelitis, or sepsis (Because the affected part is lesioned, excellent surgical results cannot be obtained.)

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 72 (Actual)
Dates: Start 2009-10-01 (Actual); Primary Completion 2012-03-31 (Actual); Study Completion 2012-03-31 (Actual)

PRIMARY OUTCOMES:
Force from femoral and tibial side to retract and bring visual field into view | intraoperatively

SECONDARY OUTCOMES:
Incision length | intraoperatively
Visual determination of the extension and flexion gap | intraoperatively

CONTACTS AND LOCATIONS:
Overall Officials: Takashi Miyamoto, MD, Principal Investigator — Osaka Medical Center
Locations (1):
- National Hospital Organization, Osaka National Hospital, Osaka, Japan